CLINICAL TRIAL: NCT01102153
Title: NSE as an Outcome Predictor of Therapeutical Hypothermia After Survived Sudden Cardiac Death
Brief Title: Neuron Specific Enolase (NSE) as Outcome Parameter of Cooling Therapy After Survived Sudden Cardiac Death
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Holger Thiele, Assistant Professor, University of Leipzig, Heart Center
Other Study IDs: COOL-NSE
Record Dates: First submitted 2010-02-08; First posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-01

CONDITIONS: Cardiac Arrest; Hypothermia
Keywords: sudden cardiac arrest; Hypothermia; Coolgard; arctic sun; neurological outcome; neuron specific enolase
MeSH Terms: conditions — Heart Arrest; Hypothermia; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Coolgard: invasive cooling
  Interventions: Device: Coolgard
- ArcticSun: non-invasive (surface) cooling
  Interventions: Device: ArcticSun

INTERVENTIONS:
Device: Coolgard — invasive cooling via femoral ICY-catheter
  Other Names: CG
  Groups: Coolgard
Device: ArcticSun — non-invasive surface cooling by saline-cooled thermo-vest
  Other Names: AS
  Groups: ArcticSun

SUMMARY:
Sudden cardiac death remains one of the major leading causes of death. Therapeutic hypothermia is a validated standard procedure to avoid or minimize cognitive deficits after cardiac arrest. To assess the efficiency of different cooling methods and further improve these methods, the investigators collected blood samples to measure the neuron specific enolase (NSE) in patients treated with invasive cooling as compared to patients treated with non-invasive cooling.

DETAILED DESCRIPTION:
Consecutive patients with restoration of spontaneous circulation after resuscitation due to sudden cardiac death were randomized to either non-invasive or invasive cooling for at least 24 hours. NSE was collected at designated time points and compared between patients treated with invasive cooling and those treated with non-invasive cooling. Neurological outcome was assessed between groups at hospital discharge and 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* ROSC after sudden cardiac death (SCA) due to VF/VT or PEA/Asystolia
* GCS 3

Exclusion Criteria:

* Non-cardiac sudden death
* Pregnancy
* Unstable circulation with high-dose inotropics
* Life-expectancy reducing concomitant illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who survived sudden cardiac arrest and where treated with cooling-therapies
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
neuron specific enolase (NSE) as a parameter for cerebral damage | 72 hours
  Blood samples were collected at predefined time-points within 72 hours to measure neuron specific enolase.

SECONDARY OUTCOMES:
neurologic outcome | 6 months
  At 6 months after cardiac arrest, the cerebral performance category score is assessed to determine neurologic outcome.
time to overall survival | one year
  At one year after cardiac arrest, overall survival of the cardiac arrest patients is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, Associate Professor, Principal Investigator — Study Chair; Undine Pittl, MD, Study Director — Study Sub-Investigator; Alexandra Schratter, MD, Study Director — Study Sub-Investigator
Locations (1):
- University of Leipzig, Heart Center, Cardiology, Leipzig, Germany

REFERENCES:
- [Background] Sulaj M, Saniova B, Drobna E, Schudichova J. Serum neuron specific enolase and malondialdehyde in patients after out-of-hospital cardiac arrest. Cell Mol Neurobiol. 2009 Sep;29(6-7):807-10. doi: 10.1007/s10571-009-9361-y. Epub 2009 Feb 25. PMID 19241153
- [Background] Shinozaki K, Oda S, Sadahiro T, Nakamura M, Hirayama Y, Abe R, Tateishi Y, Hattori N, Shimada T, Hirasawa H. S-100B and neuron-specific enolase as predictors of neurological outcome in patients after cardiac arrest and return of spontaneous circulation: a systematic review. Crit Care. 2009;13(4):R121. doi: 10.1186/cc7973. Epub 2009 Jul 22. PMID 19624826